CLINICAL TRIAL: NCT03154073
Title: Effects of Progressive Intensity Exercise Training on Glycemic Control in Older Adults Who Are at Risk for Diabetes
Brief Title: Effects of Progressive Intensity Exercise Training on Glycemic Control in Older Adults
Acronym: GLYDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-2662; F32DK116402 (NIH)
Record Dates: First submitted 2017-05-10; First posted 2017-05-15 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: PreDiabetes; Aging
Keywords: Exercise; Physical activity; Blood glucose; Sleep
MeSH Terms: conditions — Prediabetic State; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Exercise Training (Experimental): Exercise training program that will focus on engaging in ~150 minutes of moderate intensity exercise per week. Exercise will be supervised by trained staff.
  Interventions: Behavioral: Moderate Intensity Exercise Training (MOD)
- Vigorous Exercise Training (Experimental): Exercise training program that will focus on engaging in ~150 minutes of vigorous intensity exercise per week. Exercise will be supervised by trained staff.
  Interventions: Behavioral: Vigorous Intensity Exercise Training (VIG)

INTERVENTIONS:
Behavioral: Moderate Intensity Exercise Training (MOD) — For the first 4 weeks, participant will be asked to complete 3 days of exercise/week at 50-65% heart rate maximum. Sessions will last between 30-40 minutes excluding the warm-up and cool down (5-10 minutes). After 4 weeks, the MOD group will be expected to match the exercise prescription. The exercise prescription for the MOD group for weeks 5-12 will be 4 days/week, 45 min/session completed at 60-65% heart rate maximum.
  Arms: Moderate Exercise Training
Behavioral: Vigorous Intensity Exercise Training (VIG) — The exercise lead in period will be the same as the moderate intensity exercise training program. After 6 weeks, the VIG group will be expected to match the exercise prescription. The exercise prescription for the VIG for weeks 7-12 will be 4 days/week, 45 min/session completed at 80-85% heart rate maximum.
  Arms: Vigorous Exercise Training

SUMMARY:
The purpose of this study is to compare the effects of moderate versus vigorous intensity exercise training on glycemic control in older adults. Glycemic control will be assessed using an oral glucose tolerance test and continuous glucose monitors. In addition, the investigaotrs will investigate whether engaging in an exercise training program elicits changes in sedentary behavior, non-exercise physical activity, sleep, and total daily energy expenditure.

DETAILED DESCRIPTION:
Approximately 25% of older adults have type 2 diabetes mellitus, and almost 50% of older adults have prediabetes. Identifying strategies to prevent the progression of diabetes in this older adult population is imperative. One strategy that has shown promise is lifestyle modification. As adults age they also increase sedentary behavior, decrease physical activity, and have increased occurrence of sleep problems. The combination of these lifestyle factors are likely responsible for the decreases in glycemic control with aging. The American Diabetes Association recommends that prediabetic adults, including older adults, increase structured aerobic exercise and incidental (non-exercise) physical activity while decreasing sedentary behavior. It is emphasized that structured exercise is the most important of these recommendations. However, initiating an exercise routine, may unintentionally affect time spent sitting, non-exercise physical activity, and other lifestyle behaviors like sleep. These changes may attenuate or enhance the effects of exercise on glycemic control. This study will compare the effects of moderate and high intensity exercise on glycemic control, and determine whether changes in non-exercise physical activity, sitting time, and sleep are associated with the observed changes. Because of the increasing prevalence of diabetes with age, identifying the optimal exercise prescription to preserve glycemic control in older adults has important clinical implications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 to <80 years upon study entry
* Body mass index ≥25.0 to <35.0 kg/m2 as measured at the baseline screening visit
* HBA1c ≥ 5.7% to <6.5% OR Fasting Glucose ≥ 100 to <126 mg/dl as measured at the baseline screening visit.

Exclusion Criteria:

* History of metabolic, cardiac, or pulmonary disease that classifies the individual as high risk by the American College of Sports Medicine
* Participants with un-controlled hypertension and un-controlled thyroid disorders and are on medication for <3 months.
* Resting systolic blood pressure >160 mmHg or resting diastolic blood pressure >100 mmHg will be exclusionary. At the baseline screening visit, an initial resting blood pressure measurement will be attained after the participant is seated at rest for 5 minutes. Subsequent resting blood pressure measurements can be taken at the baseline screening visit up to 3 times to determine eligibility. Subsequent measurements will be taken under the same conditions as the initial measurement with a minimum of 5 minutes between readings. If more than one reading is needed to determine eligibility, the average of all readings taken will be used.
* Thyroid dysfunction, defined as an ultrasensitive thyroid stimulating hormone (TSH) <0.5 or >5.0 mU/L; volunteers with abnormal TSH values will be re-considered for participation in the study after follow-up evaluation by the PCP with initiation or adjustment of thyroid hormone replacement.
* Self-reported chronic Inflammatory Disease (e.g., rheumatoid arthritis, lupus)
* Currently taking statins, hormone replacement therapy, prescribed sleep medications, or medications that may affect heart rate response to exercise (e.g., beta blockers)
* Participating in >30 minutes of aerobic exercise/week during the past 3 months
* Inability to complete exercise test
* Sleep Apnea

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Change in Glucose Area Under the Curve (AUC) | Baseline (0 weeks), Post Intervention (12 weeks)
  Glucose will be assessed at 0, 10, 20, 30, 60, 90, 120, 180 minutes. These measurements will be used to calculate glucose AUC.
Insulin Sensitivity Index (μmol·kg^-1·min^-1·pM^-1) | Baseline (0 weeks), Post Intervention (12 weeks)
  Glucose, insulin, and c-peptide will be assessed at 0, 10, 20, 30, 60, 90, 120, 180 minutes . Height will be measured using a wall mounted stadiometer (cm). Weight will be assessed using a digital scale (kg). Collectively these measurements will be used to calculate BMI (kg/m^2). All of these measurement will be used to assess Insulin sensitivity index as determined by the regression model validated by Stumvoll.

SECONDARY OUTCOMES:
Change in Sedentary Time | Baseline (0 weeks), Post Intervention (12 weeks)
  Measured using a wearable device (min/day)
Change in Non-Exercise Physical Activity | Baseline (0 weeks), Post Intervention (12 weeks)
  Measured using a wearable device (min/day)
Change in Total Daily Energy Expenditure | Baseline (0 weeks), Post Intervention (12 weeks)
  Measured via doubly labeled water (kcals/day)
Change in Sleep Duration - 1 | Baseline (0 weeks), Post Intervention (12 weeks)
  Measured using a wearable device
Change in Sleep Duration - 2 | Baseline (0 weeks), Post Intervention (12 weeks)
  Measured using a questionnaire
Change in 24-hour Glycemic Control (glucose AUC) | Baseline (0 weeks), Post Intervention (12 weeks)
  Measured using a continuous glucose monitor (glucose AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Seth A Creasy, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No